CLINICAL TRIAL: NCT04718623
Title: Evaluation of Presepsin and Syndecan-1 as Biomarkers for Early Diagnosis and Prognosis of Sepsis Following Major Surgeries
Brief Title: Early Diagnosis and Prognosis of Postoperative Sepsis by Presepsin and Syndecan-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, hossam abousamra, specialist of anaesthesia and intensive care, Alexandria University
Other Study IDs: presepsin,syndecan-1,sepsis
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Sepsis Following A Procedure; Diagnoses, Syndromes, and Conditions
Keywords: presepsin; syndecan-1; sepsis biomarkers; following major surgeries
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous sample will be withdrawn:
  This will be assayed to all patients by enzyme-linked immune sorbent assay (ELISA) kit using double-antibody Sandwich-ELISA as the method.
  After collection of the whole blood, the blood will be left undisturbed at room temperature. This usually takes 10-20 minutes. After which the serum will be separated by centrifugation at 2000-3000 rpm for 20 minutes. Samples will be stored at -20℃ till assayed.

GROUPS / COHORTS (2):
- Sepsis group (SG): with source of infection and SOFA Score more than or equal 2
  Interventions: Diagnostic Test: Quantitative determination of serum Presepsin (sCD-14), and Syndecan-1 concentrations
- Non-Sepsis Group (NSG): with SOFA score less than 2
  Interventions: Diagnostic Test: Quantitative determination of serum Presepsin (sCD-14), and Syndecan-1 concentrations

INTERVENTIONS:
Diagnostic Test: Quantitative determination of serum Presepsin (sCD-14), and Syndecan-1 concentrations — Quantitative determination of serum Presepsin (sCD-14), and Syndecan-1 concentrations by ELISA technique

SUMMARY:
The aim of the present work is to study: Persepsin (sCD-14) and Syndecan-1 as biomarkers following major surgeries for early diagnosis and prognosis of sepsis Primary aim: early diagnosis and prognosis of sepsis Secondary aim: correlate them with SOFA and qSOFA scores.

DETAILED DESCRIPTION:
Millions of patients die around the world every year because of sepsis. 1%-2% of patients admitted to hospital and 25% of Intensive Care Units (ICU) patients suffer from sepsis. One of the most important principles of sepsis management is early diagnosis and treatment as Surviving Sepsis Campaign recommends Hour-1 bundle use.

Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection and organ dysfunction can be identified as an acute change in total Sepsis related Organ Failure Assessment (SOFA) score ≥ 2 points consequent to the infection.

The baseline SOFA score can be zero in patients not known to have pre-existing organ dysfunction. A SOFA score 2 reflects an overall mortality risk of approximately 10% in a general hospital population with suspected infection. Patients with suspected infection who are likely to have a prolonged ICU stay or die in the hospital can be promptly identified at the bedside with quick SOFA score (qSOFA) i.e. (HAT ie, Hypotension with systolic blood pressure ≤100 mm Hg, Alteration in mental status, or Tachypnea with respiratory rate ≥22/min.

Septic shock is a subset of sepsis in which underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality. Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain mean arterial blood pressure (MAP) ≥65 mm Hg and having a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation. With these criteria, hospital mortality is in excess of 40%.

As blood culture is needed to confirm diagnosis of sepsis it requires 48-72 hours to be performed, and positive rate is low. No single clinical or biological marker indicative of sepsis has been approved.

There is a need for biomarkers with a high sensitivity and specificity for early diagnosis and prognosis. They also should be positively correlating with Acute Physiology and Chronic Health Evaluation II (APACHE II) and SOFA scores.

Many known reported old biological markers as Procalcitonin (PCT), Interleukins, Pro-Vasopressin and C-Reactive Protein (CRP) have been studied and new markers were detected as Presepsin [(soluble CD14 (sCD-14)] and Syndecan-1 from Glycocalyx shedding.

One of the key molecular causes of gram-negative septicemia is a component of the outer membrane of gram-negative bacteria, lipopolysaccharide (LPS). It binds with high affinity to LPS-binding glycoproteins and activates Toll-like receptor (TLR)-4 and co-receptor cluster of differentiation 14 (CD14) expressed on monocytes/macrophages and endothelial cells to induce the secretion of proinflammatory cytokines. This is not the only main pathogenic mechanism of lipopolysaccharide (LPS). An alternative intracellular LPS-sensing pathway, bypassing TLR4, that activates caspases 4 and 5 in humans resulting in inflammasome(it is an intracellular multimeric protein complex that contains (1) a pattern recognition receptor (PRR), (2) an adaptor protein and (3) an effector enzyme (caspase), and catalyses a cellular reaction to protect against an immediate danger via cytokine secretion and cell death) induced pyroptosis has been considered to be the main pathogenic mechanism of sepsis.

Presepsin is an N-terminal fragments of 13kDa of soluble CD14 (sCD14). subtype (sCD14-ST). sCD14 is seen in plasma, and is produced by membrane-bound CD14 (mCD14) fall-off or cell secretion. Cluster of Differentiation 14 (CD14) is the receptor of lipopolysaccharide-lipopolysaccharide binding protein (LPS-LBP) complexes. CD14 has two forms: membrane-bound CD14 (mCD14) and soluble CD14 (sCD14). Presepsin is released after the binding of lipopolysaccharides (LPS) to monocytes, causing an enhanced immune response. mCD14 has a high affinity to LPS, and is mainly expressed on the cell surface of monocytes/macrophages or distributed a little bit on the cell surface of neutrophils. Two kinds of sCD14 could be detected in the plasma of healthy people at microgram level: 49KD and 55KD. sCD14 plays an important role in mediating the immune responses to LPS of CD14-negative cells such as endothelial cells and epithelial cells. sCD14 is cleaved by Cathepsin D and other proteases in plasma.

Since presepsin is produced immediately after the onset of an infection it can be detected early in the development of sepsis.its value as sepsis biomarker was shown in the diagnosis and evaluation of sepsis.

Syndecan-1 is one of components of Glycocalyx layer. This is a layer lining luminal surface of the vascular endothelium, which acts as a protective layer to maintain its permeability and a key factor in leukocyte migration and preventing intravascular coagulation.This is made of glycoproteins, proteoglycans, glycosaminoglycans and other plasma proteins especially hyaluronan and syndecans (a proteoglycan) are the principle component for its integrity.

Early pathophysiologic changes in sepsis concern the endothelium including degradation of the glycocalyx through proteinases produced by pathogens that lead to increase permeability to plasma proteins and fluids subsequently tissue edema formation and organ failure. The damaged glycocalyx layer becomes thinner and releases its components (such as syndecan-1, heparan sulfate, hyaluronan, chondroitin sulfates) into the plasma via enzymes including heparanase that cleaves the heparan sulfate and matrix metalloproteinase (MMPs) A disintegrin and metalloproteases (ADAMs). ADAM17 is inducible, cleaves syndecan-4,while ADAM10 is expressed constitutively, sheds syndecan-1 from proteoglycans. which could be used as a sepsis biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years, of either sex, after full recovery from anaesthesia and extubated, following scheduled major abdominal, abdomino-pelvic or vascular surgeries who develop an evident source of infection whether clinical, laboratory manifestation or radiological signs of infection and/or criteria of quick SOFA (qSOFA) after admission to ICU will be included in the study.

Exclusion Criteria:

1. Patients aged <18 years old.
2. Patients with terminal stage of malignancy of any type.
3. Immune-compromised patients e.g., on immune-suppressive therapy, acquired immunodeficiency syndrome
4. Patients with end-stage liver or renal disease.
5. Patients with existing infection before surgery.
6. Patients with emergency surgeries.
7. Pregnancy.
8. Chronic inflammatory disorders e.g., sarcoidosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged ≥18 years, of either sex, after full recovery from anaesthesia and extubated, following scheduled major abdominal, abdomino-pelvic or vascular surgeries who develop an evident source of infection whether clinical, laboratory manifestation or radiological signs of infection and/or criteria of quick SOFA (qSOFA) after admission to ICU will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate Presepsin (sCD-14) and Syndecan-1 as biomarkers following major surgeries for early diagnosis and prognosis of sepsis | baseline
  measure quantitative concentrations of Persepsin (sCD-14) and Syndecan-1 as biomarkers for early diagnosis and predict outcome

SECONDARY OUTCOMES:
correlate Persepsin (sCD-14) and Syndecan-1 with SOFA and qSOFA scores. | baseline
  evaluation of level of Persepsin (sCD-14) and Syndecan-1 with SOFA and qSOFA scores to find if there is relationship between them

CONTACTS AND LOCATIONS:
Overall Officials: Hesham F Shaaban, Prof, Study Director — University of Alexandria; Rania Sh Swelem, Prof, Study Director — University of Alexandria; Hussien W Hussein, PHD, Study Director — University of Alexandria

REFERENCES:
- [Background] Napolitano LM. Sepsis 2018: Definitions and Guideline Changes. Surg Infect (Larchmt). 2018 Feb/Mar;19(2):117-125. doi: 10.1089/sur.2017.278. PMID 29447109
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Soong J, Soni N. Sepsis: recognition and treatment. Clin Med (Lond). 2012 Jun;12(3):276-80. doi: 10.7861/clinmedicine.12-3-276. No abstract available. PMID 22783783
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Background] Lehman KD. Update: Surviving Sepsis Campaign recommends Hour-1 bundle use. Nurse Pract. 2019 Apr;44(4):10. doi: 10.1097/01.NPR.0000554123.08252.ae. No abstract available. PMID 30768497
- [Background] Cortes-Puch I, Hartog CS. Opening the Debate on the New Sepsis Definition Change Is Not Necessarily Progress: Revision of the Sepsis Definition Should Be Based on New Scientific Insights. Am J Respir Crit Care Med. 2016 Jul 1;194(1):16-8. doi: 10.1164/rccm.201604-0734ED. No abstract available. PMID 27166972
- [Background] Goulden R, Hoyle MC, Monis J, Railton D, Riley V, Martin P, Martina R, Nsutebu E. qSOFA, SIRS and NEWS for predicting inhospital mortality and ICU admission in emergency admissions treated as sepsis. Emerg Med J. 2018 Jun;35(6):345-349. doi: 10.1136/emermed-2017-207120. Epub 2018 Feb 21. PMID 29467173
- [Background] Wentowski C, Mewada N, Nielsen ND. Sepsis in 2018: a review. Anaesth. Intensive Care Med. 2019;20(1):6-13
- [Background] Lu YH, Liu L, Qiu XH, Yu Q, Yang Y, Qiu HB. Effect of early goal directed therapy on tissue perfusion in patients with septic shock. World J Emerg Med. 2013;4(2):117-22. doi: 10.5847/wjem.j.issn.1920-8642.2013.02.006. PMID 25215104
- [Background] Hung SK, Lan HM, Han ST, Wu CC, Chen KF. Current Evidence and Limitation of Biomarkers for Detecting Sepsis and Systemic Infection. Biomedicines. 2020 Nov 12;8(11):494. doi: 10.3390/biomedicines8110494. PMID 33198109
- [Background] Caramore TJ, La Rocca R, Richards E. Does procalcitonin predict sepsis in critically ill patients? EBP. 2019;22(1):14-5.
- [Background] Guignant C, Voirin N, Venet F, Poitevin F, Malcus C, Bohe J, Lepape A, Monneret G. Assessment of pro-vasopressin and pro-adrenomedullin as predictors of 28-day mortality in septic shock patients. Intensive Care Med. 2009 Nov;35(11):1859-67. doi: 10.1007/s00134-009-1610-5. Epub 2009 Aug 7. PMID 19662382
- [Background] Povoa P. C-reactive protein: a valuable marker of sepsis. Intensive Care Med. 2002 Mar;28(3):235-43. doi: 10.1007/s00134-002-1209-6. Epub 2002 Feb 6. No abstract available. PMID 11904651
- [Background] Venugopalan DP, Pillai G, Krishnan S. Diagnostic Value and Prognostic Use of Presepsin Versus Procalcitonin in Sepsis. Cureus. 2019 Jul 16;11(7):e5151. doi: 10.7759/cureus.5151. PMID 31523578
- [Background] Uchimido R, Schmidt EP, Shapiro NI. The glycocalyx: a novel diagnostic and therapeutic target in sepsis. Crit Care. 2019 Jan 17;23(1):16. doi: 10.1186/s13054-018-2292-6. PMID 30654825
- [Background] Holzmann MS, Winkler MS, Strunden MS, Izbicki JR, Schoen G, Greiwe G, Pinnschmidt HO, Poppe A, Saugel B, Daum G, Goetz AE, Heckel K. Syndecan-1 as a biomarker for sepsis survival after major abdominal surgery. Biomark Med. 2018 Feb;12(2):119-127. doi: 10.2217/bmm-2017-0231. Epub 2018 Jan 12. PMID 29327601
- [Background] Amin J, Boche D, Rakic S. What do we know about the inflammasome in humans? Brain Pathol. 2017 Mar;27(2):192-204. doi: 10.1111/bpa.12479. PMID 27997042
- [Background] Goligorsky MS, Sun D. Glycocalyx in Endotoxemia and Sepsis. Am J Pathol. 2020 Apr;190(4):791-798. doi: 10.1016/j.ajpath.2019.06.017. Epub 2020 Feb 6. PMID 32035882
- [Background] Grunwald U, Kruger C, Westermann J, Lukowsky A, Ehlers M, Schutt C. An enzyme-linked immunosorbent assay for the quantification of solubilized CD14 in biological fluids. J Immunol Methods. 1992 Nov 5;155(2):225-32. doi: 10.1016/0022-1759(92)90289-6. PMID 1385535
- [Background] Landmann R, Zimmerli W, Sansano S, Link S, Hahn A, Glauser MP, Calandra T. Increased circulating soluble CD14 is associated with high mortality in gram-negative septic shock. J Infect Dis. 1995 Mar;171(3):639-44. doi: 10.1093/infdis/171.3.639. PMID 7533199
- [Background] Colbert JF, Schmidt EP. Endothelial and Microcirculatory Function and Dysfunction in Sepsis. Clin Chest Med. 2016 Jun;37(2):263-75. doi: 10.1016/j.ccm.2016.01.009. Epub 2016 Mar 4. PMID 27229643
- [Background] Mussap M, Noto A, Fravega M, Fanos V. Soluble CD14 subtype presepsin (sCD14-ST) and lipopolysaccharide binding protein (LBP) in neonatal sepsis: new clinical and analytical perspectives for two old biomarkers. J Matern Fetal Neonatal Med. 2011 Oct;24 Suppl 2:12-4. doi: 10.3109/14767058.2011.601923. PMID 21740312
- [Background] Shirakawa K, Naitou K, Hirose J, Takahashi T, Furusako S. Presepsin (sCD14-ST): development and evaluation of one-step ELISA with a new standard that is similar to the form of presepsin in septic patients. Clin Chem Lab Med. 2011 May;49(5):937-9. doi: 10.1515/CCLM.2011.145. Epub 2011 Feb 11. No abstract available. PMID 21345045
- [Background] Kondo Y, Umemura Y, Hayashida K, Hara Y, Aihara M, Yamakawa K. Diagnostic value of procalcitonin and presepsin for sepsis in critically ill adult patients: a systematic review and meta-analysis. J Intensive Care. 2019 Apr 15;7:22. doi: 10.1186/s40560-019-0374-4. eCollection 2019. PMID 31016020
- [Background] Aliu-Bejta A, Atelj A, Kurshumliu M, Dreshaj S, Barsic B. Presepsin values as markers of severity of sepsis. Int J Infect Dis. 2020 Jun;95:1-7. doi: 10.1016/j.ijid.2020.03.057. Epub 2020 Apr 3. PMID 32251795
- [Background] Bosch F, Schallhorn S, Miksch RC, Chaudry IH, Faist E, Werner J, Angele MK, Pratschke S. The Prognostic Value of Presepsin for Sepsis in Abdominal Surgery: A Prospective Study. Shock. 2020 Jul;54(1):56-61. doi: 10.1097/SHK.0000000000001479. PMID 31743301
- [Background] Yang Y, Schmidt EP. The endothelial glycocalyx: an important regulator of the pulmonary vascular barrier. Tissue Barriers. 2013 Jan 1;1(1):e23494. doi: 10.4161/tisb.23494. PMID 24073386
- [Background] Reitsma S, Slaaf DW, Vink H, van Zandvoort MA, oude Egbrink MG. The endothelial glycocalyx: composition, functions, and visualization. Pflugers Arch. 2007 Jun;454(3):345-59. doi: 10.1007/s00424-007-0212-8. Epub 2007 Jan 26. PMID 17256154
- [Background] Chelazzi C, Villa G, Mancinelli P, De Gaudio AR, Adembri C. Glycocalyx and sepsis-induced alterations in vascular permeability. Crit Care. 2015 Jan 28;19(1):26. doi: 10.1186/s13054-015-0741-z. PMID 25887223
- [Background] Fleck A, Raines G, Hawker F, Trotter J, Wallace PI, Ledingham IM, Calman KC. Increased vascular permeability: a major cause of hypoalbuminaemia in disease and injury. Lancet. 1985 Apr 6;1(8432):781-4. doi: 10.1016/s0140-6736(85)91447-3. PMID 2858667
- [Background] Chappell D, Jacob M, Rehm M, Stoeckelhuber M, Welsch U, Conzen P, Becker BF. Heparinase selectively sheds heparan sulphate from the endothelial glycocalyx. Biol Chem. 2008 Jan;389(1):79-82. doi: 10.1515/BC.2008.005. PMID 18095872
- [Background] Mishra HK, Ma J, Walcheck B. Ectodomain Shedding by ADAM17: Its Role in Neutrophil Recruitment and the Impairment of This Process during Sepsis. Front Cell Infect Microbiol. 2017 Apr 25;7:138. doi: 10.3389/fcimb.2017.00138. eCollection 2017. PMID 28487846
- [Background] Karakike E, Kyriazopoulou E, Tsangaris I, Routsi C, Vincent JL, Giamarellos-Bourboulis EJ. The early change of SOFA score as a prognostic marker of 28-day sepsis mortality: analysis through a derivation and a validation cohort. Crit Care. 2019 Nov 29;23(1):387. doi: 10.1186/s13054-019-2665-5. PMID 31783881
- [Background] Raith EP, Udy AA, Bailey M, McGloughlin S, MacIsaac C, Bellomo R, Pilcher DV; Australian and New Zealand Intensive Care Society (ANZICS) Centre for Outcomes and Resource Evaluation (CORE). Prognostic Accuracy of the SOFA Score, SIRS Criteria, and qSOFA Score for In-Hospital Mortality Among Adults With Suspected Infection Admitted to the Intensive Care Unit. JAMA. 2017 Jan 17;317(3):290-300. doi: 10.1001/jama.2016.20328. PMID 28114553
- [Background] Ladakis C, Myrianthefs P, Karabinis A, Karatzas G, Dosios T, Fildissis G, Gogas J, Baltopoulos G. Central venous and mixed venous oxygen saturation in critically ill patients. Respiration. 2001;68(3):279-85. doi: 10.1159/000050511. PMID 11416249
- [Background] Dueck MH, Klimek M, Appenrodt S, Weigand C, Boerner U. Trends but not individual values of central venous oxygen saturation agree with mixed venous oxygen saturation during varying hemodynamic conditions. Anesthesiology. 2005 Aug;103(2):249-57. doi: 10.1097/00000542-200508000-00007. PMID 16052106
- [Background] Berridge JC. Influence of cardiac output on the correlation between mixed venous and central venous oxygen saturation. Br J Anaesth. 1992 Oct;69(4):409-10. doi: 10.1093/bja/69.4.409. PMID 1419454
- [Background] Tahvanainen J, Meretoja O, Nikki P. Can central venous blood replace mixed venous blood samples? Crit Care Med. 1982 Nov;10(11):758-61. doi: 10.1097/00003246-198211000-00012. PMID 7140317